CLINICAL TRIAL: NCT01353560
Title: Use and Effectiveness of a Model Integrative Care Clinic in an Academic Hospital: Study 1-Survey
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Julie E. Buring, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: 1R01AT005065-01A1-1; 1R01AT005065-01A1 (NIH)
Record Dates: First submitted 2011-05-12; First posted 2011-05-13 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Medical Care
Keywords: integrative medicine; barriers to utilization; communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- New patients of Osher Clinical Center

SUMMARY:
Despite widespread and growing popularity of complementary and alternative medicine (CAM) in the US, there currently exist significant gaps in our knowledge regarding CAM use, clinical effectiveness, safety and cost- effectiveness. With previous funding support from NCCAM, the Harvard Medical School (HMS) Osher Research Center established and trained a multidisciplinary integrative team of CAM and conventional providers to work collaboratively to provide state-of-the-art "integrative care" in a coordinated and individualized fashion. The Osher Integrative Care Center (OCC) was opened in fall 2007, physically located within the Ambulatory Care Center of the Brigham and Women's Hospital (BWH) at 850 Boylston Street in Chestnut Hill, MA. The focus of this survey study is to characterize the decision-making process of both patients and conventional providers with respect to communication about and referral to an integrative care team in an academic hospital outpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* New patient coming into Osher Clinical Center for any medical reason.
* Physician affiliated with any of included division/department (see above).

Exclusion Criteria:

* Patient has been seen at Osher Clinical Center within past 3 months for any reason.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. All new patients coming into the Osher Clinical Center (OCC) for any medical reason.
  2. All physicians in the 5 included departments/divisions (Women's Health, Orthopedics, Obstetrics and Gynecology, General Medicine, and Rheumatology) are eligible to participate in the survey. Other BWH physicians whom OCC patients have identified as their referring doctors and given us permission to contact, will also be eligible to participate in the survey.
Sampling Method: Non-Probability Sample
Enrollment: 1509 (Actual)
Dates: Start 2011-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Characterization of decision-making process for patients of CAM therapies and conventional providers | 3.5 years
  Surveys will be sent to: 1) 1500 consecutive new patients seen at the OCC over 3.5 years, to characterize the chief complaints; their medical history; referral sources; communication with their physicians; barriers to use of CAM; views regarding and previous use of CAM; and expectations for CAM therapy as adjuncts to their conventional care; 2) 300 BWH physicians from five divisions (Women's Health, Orthopedics, Obstetrics and Gynecology, General Medicine, and Rheumatology) most likely to refer to the OCC, to assess their use of, feelings about, and knowledge of CAM.

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Buring, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Osher Clinical Center at Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States